CLINICAL TRIAL: NCT07404449
Title: Effects of Sex-Speciffic Compound Food Supplements on Changes in Biomarkers and Epigenetic Changes Associated With Longevity
Brief Title: Sex-Speciffic Longevity Food Supplements
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: Biostile d.o.o. (Unknown)
Responsible Party: Principal Investigator, Nina Mohorko, Associate Professor, University of Primorska
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DOLGOZIVOST
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Aging
Keywords: biological age; food supplement; longevity

STUDY DESIGN:
Intervention Model Description: Double blind intervention study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Female longevity food supplement (Experimental): 6-month daily consumption of 2 capsules of female food supplement in the morning.
  Interventions: Dietary Supplement: compound food supplements - female specific
- Female placebo (Placebo Comparator): 6-month daily consumption of 2 capsules of maltodextrin in the morning.
  Interventions: Dietary Supplement: Placebo
- Male longevity food supplement (Experimental): 6-month daily consumption of 2 capsules of male food supplement in the morning.
  Interventions: Dietary Supplement: compound food supplements - male specific
- Male placebo (Placebo Comparator): 6-month daily consumption of 2 capsules of maltodextrin in the morning.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: compound food supplements - female specific — 2 capsules per day at breakfast with glass of water for 6 months.
  Arms: Female longevity food supplement
Dietary Supplement: compound food supplements - male specific — 2 capsules per day at breakfast with glass of water for 6 months.
  Arms: Male longevity food supplement
Dietary Supplement: Placebo — 2 capsules per day at breakfast with glass of water for 6 months.
  Arms: Female placebo; Male placebo

SUMMARY:
The use of food supplements with the aim of increasing longevity in the general population is rapidly increasing, while high-quality clinical evidence on the efficacy of comprehensive formulations and their impact on biomarkers of aging is lacking. We will perform a double-blind, placebo-controlled, randomized clinical trial of a selected sex-specific dietary supplement in relation to longevity in a selected population of healthy adults of both sexes between the ages of 50 and 70.

The main questions it answers are:

Does the 6-month use of the longevity supplement impacts the 6-months change in different markers for measuring biological age compared to placebo?

Our study will involve 60 subjects, of whom 30 will consume the sex-specific longevity food supplements and 30 will consume a placebo.

The study will last 6 months. The subjects will visit the Faculty four times: at the beginning of the study (background measurement), after one, three and six months of consuming the dietary supplement or placebo.

At each visit, subjects will undergo anthropometric measurements, blood pressure measurements, and blood samples will be taken to determine baseline haematocrite, albumin, creatinine, alcaline phosphatase, lipid profile, glucose concentration, inflammatory parameters, antioxidant potential, inflammatory markers, liver enzymes, and expression of genes for autophagy and oxidative stress. Subjects will also complete 3-day food diaries and questionnaires on general health, physical activity, and quality of sleep and life.

On baseline and final (six months) measurements resting metabolic rate, DXA body composition measurements will be performed and saliva samples will be obtained for DNA methilation determination.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 22 kg/m2 and 30 kg/m2
* Postmenopausal women (at least 12 months without menstruation)
* Healthy individuals, without risk of chronic non-communicable diseases
* Signed written informed consent

Exclusion Criteria:

1. Acute and chronic diseases (cardiovascular diseases, diabetes, neurodegenerative diseases, gastrointestinal diseases)
2. Patients with serious clinical conditions such as cancer, severe infections, severe psychiatric disorders, autoimmune diseases, inflammatory diseases
3. BMI less than 22 kg/m2 and greater than 30 kg/m2
4. Celiac disease or gluten intolerance
5. Presence of implants, devices or other foreign materials in the measurement area
6. Smoking
7. Atypical sleep patterns
8. Use of dietary supplements and medications
9. Extreme physical activity
10. Excessive alcohol consumption (more than one drink per day for women, more than two drinks per day for men)

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Albumin | From enrollment to the end of last measurement at 6 months.
  Albumin levels will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Creatinine | From enrollment to the end of last measurement at 6 months.
  Creatinine levels will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Glucose | From enrollment to the end of last measurement at 6 months.
  Glucose levels will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
CRP | From enrollment to the end of last measurement at 6 months.
  CRP levels will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Lymphocyte percent | From enrollment to the end of last measurement at 6 months.
  Lymphocyte percent will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Mean cell volume | From enrollment to the end of last measurement at 6 months.
  Mean cell volume will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Red cell distribution width | From enrollment to the end of last measurement at 6 months.
  Red cell distribution width will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Alcaline phosphatase | From enrollment to the end of last measurement at 6 months.
  Alcaline phosphatase will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
White blood cell count | From enrollment to the end of last measurement at 6 months.
  White blood cell count will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
PhenoAge | From enrollment to the end of last measurement at 6 months.
  PhenoAge will be calculated from albumin, creatinine, glucose, lymphocyte percent, mean cell volume, red cell distribution width, alcaline phosphatase, white blood cell count and cronological age at baseline, after 1, 3 and 6 months of daily dietary supplements use (according to Ruan et al, 2023).
DNA methylation | From enrollment to the end of last measurement at 6 months.
  DNA methylation will be measured from saliva at baseline and 6 months of daily dietary supplements use.
Horvath epigenetic age | From enrollment to the end of last measurement at 6 months.
  Horvath epigenetic age will be determined from saliva DNA methylation data (according to Horvath & Raj, 2018) at baseline and 6 months of daily dietary supplements use..

SECONDARY OUTCOMES:
Total cholesterol | From enrollment to the end of last measurement at 6 months.
  Total cholesterol levels will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
LDL cholestorol | From enrollment to the end of last measurement at 6 months.
  LDL cholesterol levels will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
HDL cholesterol | From enrollment to the end of last measurement at 6 months.
  HDL cholesterol levels will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Triacylglycerols | From enrollment to the end of last measurement at 6 months.
  Triacylglycerols levels will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Antioxidant potential | From enrollment to the end of last measurement at 6 months.
  Antioxidant potential will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Aspartate aminotransferase (AST) | From enrollment to the end of last measurement at 6 months.
  AST will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Alanine aminotransferase (ALT) | From enrollment to the end of last measurement at 6 months.
  ALT will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Interleukine-6 (IL-6) | From enrollment to the end of last measurement at 6 months.
  IL-6 will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Tumor necrosis factor alpha (TNF-alpha) | From enrollment to the end of last measurement at 6 months.
  TNF-alpha will be measured from venous blood at baseline, after 1, 3 and 6 months of daily dietary supplements use.
NAD+/NADH | From enrollment to the end of last measurement at 6 months.
  NAD+/NADH ratio will be measured from venous blood at baseline and 6 months of daily dietary supplements use.
Sleep quality | From enrollment to the end of last measurement at 6 months.
  Sleep quality will be assessed with THe Pittsburgh Sleep Quality Index questionnaire (Buysse et al., 1989) at baseline, after 1, 3 and 6 months of daily dietary supplements use.
World Health Organization-FIve Well.Being Index | From enrollment to the end of last measurement at 6 months.
  Quality of life will be assessed with World Health Organization-FIve Well.Being Index (WHO5 questionnaire, Slovenian translation, WHO, 2024) at baseline, after 1, 3 and 6 months of daily dietary supplements use.
BMAL1 gene expression | From enrollment to the end of last measurement at 6 months.
  BMAL1 gene expression will be determined from Lymphocyte fraction at baseline and 6 months of daily dietary supplements use.
ATG1 gene expression | From enrollment to the end of last measurement at 6 months.
  ATG1 gene expression will be determined from Lymphocyte fraction at baseline and 6 months of daily dietary supplements use.
SD1 gene expression | From enrollment to the end of last measurement at 6 months.
  SD1 gene expression will be determined from Lymphocyte fraction at baseline and 6 months of daily dietary supplements use.
mTOR gene rxpression | From enrollment to the end of last measurement at 6 months.
  mTOR gene expression will be determined from Lymphocyte fraction at baseline and 6 months of daily dietary supplements use.
SIRT1 gene expression | From enrollment to the end of last measurement at 6 months.
  SIRT1 gene expression will be determined from Lymphocyte fraction at baseline and 6 months of daily dietary supplements use.
glutation reductase gene expression | From enrollment to the end of last measurement at 6 months.
  Glutation reductase gene expression will be determined from Lymphocyte fraction at baseline and 6 months of daily dietary supplements use.

OTHER OUTCOMES:
Anthropometric assessment | From enrollment to the end of last measurement at 6 months.
  Body mass and body composition will be measured with body scale and bioimpedance analysator at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Blood pressure | From enrollment to the end of last measurement at 6 months.
  Blood pressure will be measured at baseline, after 1, 3 and 6 months of daily dietary supplements use.
Physical activity level | From enrollment to the end of last measurement at 6 months.
  Physical activity level will be assessed with IPAQ questionnaire at baseline, after 1, 3 and 6 months of daily dietary supplements use.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Petelin, PhD, Principal Investigator — University of Primorska, Faculty of Health Sciences
Locations (1):
- University pf Primorska, Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kyle UG, Bosaeus I, De Lorenzo AD, Deurenberg P, Elia M, Gomez JM, Heitmann BL, Kent-Smith L, Melchior JC, Pirlich M, Scharfetter H, Schols AM, Pichard C; Composition of the ESPEN Working Group. Bioelectrical impedance analysis--part I: review of principles and methods. Clin Nutr. 2004 Oct;23(5):1226-43. doi: 10.1016/j.clnu.2004.06.004. PMID 15380917
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Horvath S. DNA methylation age of human tissues and cell types. Genome Biol. 2013;14(10):R115. doi: 10.1186/gb-2013-14-10-r115. PMID 24138928
- [Background] Horvath S, Raj K. DNA methylation-based biomarkers and the epigenetic clock theory of ageing. Nat Rev Genet. 2018 Jun;19(6):371-384. doi: 10.1038/s41576-018-0004-3. PMID 29643443
- [Background] Ruan Z, Li D, Huang D, Liang M, Xu Y, Qiu Z, Chen X. Relationship between an ageing measure and chronic obstructive pulmonary disease, lung function: a cross-sectional study of NHANES, 2007-2010. BMJ Open. 2023 Nov 2;13(11):e076746. doi: 10.1136/bmjopen-2023-076746. PMID 37918922
- See also: WHO5 Slovenian translation — https://cdn.who.int/media/docs/default-source/mental-health/five-well-being-index-(who-5)/who-5_slovenian.pdf?sfvrsn=f9adb3c4_3